CLINICAL TRIAL: NCT04033341
Title: Disposition of [14C]-LY3214996 Following Oral Administration in Healthy Male Subjects
Brief Title: A Study of LY3214996 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17199; I8S-MC-JUAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — LY3214996

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3214996 + [14C]-LY3214996 (Experimental): A single dose of LY3214996 and [14C]-LY3214996 administered orally.
  Interventions: Drug: LY3214996; Drug: [14C]-LY3214996

INTERVENTIONS:
Drug: LY3214996 — Administered orally
Drug: [14C]-LY3214996 — Administered orally

SUMMARY:
The main purpose of this study is to measure how much of the study drug gets into the bloodstream and how long it takes the body to get rid of it. This study will involve a single dose of 14C radiolabelled LY3214996. This means that a radioactive substance, C14, will be incorporated into the study drug. The purposes are to investigate the study drug and its breakdown products and to find out how much of these pass from blood into urine and feces. The study will last up to six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Overtly health males
* Body mass index (BMI) of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive

Exclusion Criteria:

* Females
* Male participants sexually active with a pregnant partner
* Are currently enrolled in a clinical study or have participated, within the last 30 days, in a clinical study
* Have participated in a radiolabeled drug study within the previous 4 months
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders
* Have a history of Gilbert's syndrome
* Have history or presence of psychiatric disorders
* Show evidence of human immunodeficiency virus (HIV) infection
* Show evidence of hepatitis C
* Show evidence of hepatitis B

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Urinary Excretion of LY3214996 Radioactivity Over Time Expressed As A Percentage of the Total Radioactive Dose Administered | Baseline through Day 8 after administration of study drug
  Urinary Excretion of LY3214996 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Fecal Excretion of LY3214996 Radioactivity Over Time Expressed As A Percentage of the Total Radioactive Dose Administered | Baseline through Day 8 after administration of study drug
  Fecal Excretion of LY3214996 Radioactivity Over Time Expressed As A Percentage of the Total Radioactive Dose Administered

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3214996 | Predose through Day 8 after administration of study drug
  PK: Cmax of LY3214996
PK: Area Under the Concentration Time Curve From Time Zero to Infinity (AUC[0-∞]) of LY3214996 | Predose through Day 8 after administration of study drug
  PK: AUC(0-∞) of LY3214996
Total Number of Metabolites of LY3214996 | Baseline through 48 hours after administration of study drug
  Total Number of Metabolites of LY3214996

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No